CLINICAL TRIAL: NCT03999632
Title: Effects of Aquatic Plant Protein Source Wolffia Globosa (Mankai) on Weight Loss, Cardiometabolic State, and Patient's Satisfaction During the Preoperative Dietary Intervention Period in Patients Undergoing Bariatric Surgery.
Brief Title: Effects of Wolffia Globosa (Mankai) in Patients Undergoing Bariatric Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Clinic Florida (Other)
Responsible Party: Principal Investigator, Emanuele LoMenzo, Principal Investigator, Director Department of Research,, Cleveland Clinic Florida
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FLA 18-070
Record Dates: First submitted 2019-04-17; First posted 2019-06-27 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Bariatric Surgery Candidate; Diet Modification
Keywords: Bariatric surgery; Sleeve gastrectomy; Preoperative diet; Hepatic steatosis; Wolffia Globosa; Hyperglycemia
MeSH Terms: conditions — Fatty Liver; Hyperglycemia | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mankai Group (Experimental): The pre-operative liquid diet will be started two weeks before surgery date for both groups. During the first week patients in group A (Wolffia Globosa) will be allowed to have two meals a day and one protein shake (Wolffia Globosa) of 16 oz. Each meal will consist of 3-5 oz of lean protein (Chicken, turkey or fish) and one cup of vegetables or salad. During the second week, patients will drink one protein shake of 16 oz (Wolffia Globosa) as a meal replacement, three times per day and will not be allowed to eat solid food. Patients will also be allowed to Drink clear liquids in between protein shakes.
  Interventions: Other: Dietary modification with introduction of Mankai
- Control Group (No Intervention): The pre-operative liquid diet will be started two weeks before surgery date for both groups. During the first week patients in group B (Control) will be allowed to have two meals a day and one protein shake (Control) of 16 oz. Each meal will consist of 3-5 oz of lean protein (Chicken, turkey or fish) and one cup of vegetables or salad. During the second week, patients will drink one protein shake of 16 oz (Control) as a meal replacement, three times per day and will not be allowed to eat solid food. Patients will also be allowed to Drink clear liquids in between protein shakes.

INTERVENTIONS:
Other: Dietary modification with introduction of Mankai — Substituting the standard high protein, low carbohydrate preoperative shake during the preoperative liquid diet with Wolffia Globosa (Mankai) shake consisting of 16 oz of skim milk + 1 frozen cube of Wolffia Globosa (Mankai) +/- sugar substitute.
  Arms: Mankai Group

SUMMARY:
Candidates to bariatric surgery at The Bariatric and Metabolic Institute at Cleveland Clinic Florida are prescribed a high protein liquid diet for two weeks preoperatively and 2 weeks postoperatively. Whether Wolffia Globosa (Mankai), a plant based wholesome food, can serve as a natural alternative to liquid diet during the 2 week pre-operation and 2 weeks postoperation liquid based diet, is unknown.

The investigators aim to address the effect of daily Wolffia Globosa (Mankai) administration on morbid/severely-obese patients during the 2 week pre-operative period and 2 weeks postoperatively as compared to iso protein-iso caloric shake source on the following parameters

DETAILED DESCRIPTION:
This study is a prospective study involving patients selected for elective surgery. Patients undergoing bariatric surgery will be enrolled in this study and have several parameters checked as explained below. Patients selected and consented for elective bariatric surgery will be recruited in the Bariatric and Metabolic Institute to participate in this study and will undergo standard of care. The investigators will enroll approximately 120 candidates during a 6 months (~5 a week) period. Patients will be randomized to the A. control group: 3 traditional shakes or B. intervention group: 2 traditional shakes and 1 daily administration of substituting iso-protein green Wolffia Globosa (Mankai) Shake (4 frozen cubes of Wolffia Globosa (Mankai) equal to 20 grams of dry Wolffia Globosa (Mankai). Each shake will provide equivalent carbohydrate, calories and protein levels from the respective source. As part of our routine pre and postoperative screening and follow up protocol, the investigators will collect anthropometric and clinical data on all patients, including standard of care blood samples collected at 2 weeks pre operatively, surgery day and at 2 months postoperatively

ELIGIBILITY:
Inclusion Criteria:

• Patients that will undergo sleeve gastrectomy.

Exclusion Criteria:

* Age below 18 years
* American Society of Anesthesiologist (ASA) class IV or V
* Patients using Vitamin-K antagonists
* Patients with documented coagulopathies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Patient's Satiety with Wolffia Globosa (Mankai) shake measured with a QUALITY OF ALIMENTATION QUESTIONNAIRE | 2 weeks
  QUALITY OF ALIMENTATION QUESTIONNAIRE is a questionnaire with 1 open ended question, 4 yes/no questions, and three 0-5 questions with 5 being the highest level
Glucose control in patients with previous Type 2 Diabetes Mellitus diagnosis by fasting glucose and Hgb A1c | 2 weeks
  Glucose control in patients with previous Type 2 Diabetes Mellitus diagnosis (T2DM). measure by fasting glucose and Hgb A1c
Patient's liking with Wolffia Globosa (Mankai) shake measured with a questionnaire | 2 weeks
  Patient's liking with Wolffia Globosa (Mankai) shake. measured with a questionnaire
Patient's tolerance with Wolffia Globosa (Mankai) shake. measured with a questionnaire | 2 weeks
  QUALITY OF ALIMENTATION QUESTIONNAIRE is a questionnaire with 1 open ended question, 4 yes/no questions, and three 0-5 questions with 5 being the highest level
Patient's compliance with Wolffia Globosa (Mankai) shake. measured with a questionnaire | 2 weeks
  QUALITY OF ALIMENTATION QUESTIONNAIRE is a questionnaire with 1 open ended question, 4 yes/no questions, and three 0-5 questions with 5 being the highest level

SECONDARY OUTCOMES:
Metabolic and nutritional effects of Wolffia Globosa (Mankai) in patients undergoing bariatric surgery by serum measurements | 2.5 months
  Serum levels of the common nutritional parameters will be checked before and after the intervention
Adverse effect by patient report and clinical follow up | 2.5 months
  Adverse effect patient report and clinical follow up
Fat% (via Bioelectrical Impedance) | 2.5 months
  Fat% (via Bioelectrical Impedance)
Fatty liver infiltration by Ultrasound | 2.5 months
  Fatty liver infiltration by Ultrasound
Patient's adherence by food diary | 2.5 months
  Patient's adherence by food diary
Satisfaction of Patients by specific questionnaire | 2.5 months
  Satisfaction of Patients. by specific questionnaire
Free Fat Mass (via Bioelectrical Impedance) | 2.5 months
  Free Fat Mass (via Bioelectrical Impedance)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Lo Menzo, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Confidentiality and Privacy:
  Information about study subjects will be kept confidential and managed according to the Health Insurance Portability and Accountability Act of 1996 (HIPAA).
  Source Documents:
  Source data will include the electronic health record for patient demographics, vitals, and basic laboratory results. Dictated operative notes will be maintained within the EHR as well. Lab results of inflammatory markers will be kept out of the EHR and kept in a secure file on the Cleveland Clinic server.
  Records Retention:
  The investigators will retain study essential documents for at least six years after completion of the research and are accessible for inspection by authorized representatives at reasonable times and in a reasonable manner.

REFERENCES:
- [Background] Gilani GS, Cockell KA, Sepehr E. Effects of antinutritional factors on protein digestibility and amino acid availability in foods. J AOAC Int. 2005 May-Jun;88(3):967-87. PMID 16001874
- [Background] Sarwar Gilani G, Wu Xiao C, Cockell KA. Impact of antinutritional factors in food proteins on the digestibility of protein and the bioavailability of amino acids and on protein quality. Br J Nutr. 2012 Aug;108 Suppl 2:S315-32. doi: 10.1017/S0007114512002371. PMID 23107545
- [Background] Pan A, Sun Q, Bernstein AM, Schulze MB, Manson JE, Stampfer MJ, Willett WC, Hu FB. Red meat consumption and mortality: results from 2 prospective cohort studies. Arch Intern Med. 2012 Apr 9;172(7):555-63. doi: 10.1001/archinternmed.2011.2287. Epub 2012 Mar 12. PMID 22412075
- [Background] Chalvon-Demersay T, Azzout-Marniche D, Arfsten J, Egli L, Gaudichon C, Karagounis LG, Tome D. A Systematic Review of the Effects of Plant Compared with Animal Protein Sources on Features of Metabolic Syndrome. J Nutr. 2017 Mar;147(3):281-292. doi: 10.3945/jn.116.239574. Epub 2017 Jan 25. PMID 28122929
- [Background] Micha R, Wallace SK, Mozaffarian D. Red and processed meat consumption and risk of incident coronary heart disease, stroke, and diabetes mellitus: a systematic review and meta-analysis. Circulation. 2010 Jun 1;121(21):2271-83. doi: 10.1161/CIRCULATIONAHA.109.924977. Epub 2010 May 17. PMID 20479151
- [Background] Wang X, Lin X, Ouyang YY, Liu J, Zhao G, Pan A, Hu FB. Red and processed meat consumption and mortality: dose-response meta-analysis of prospective cohort studies. Public Health Nutr. 2016 Apr;19(5):893-905. doi: 10.1017/S1368980015002062. Epub 2015 Jul 6. PMID 26143683
- [Background] Pan A, Sun Q, Bernstein AM, Schulze MB, Manson JE, Willett WC, Hu FB. Red meat consumption and risk of type 2 diabetes: 3 cohorts of US adults and an updated meta-analysis. Am J Clin Nutr. 2011 Oct;94(4):1088-96. doi: 10.3945/ajcn.111.018978. Epub 2011 Aug 10. PMID 21831992
- [Background] Malik VS, Li Y, Tobias DK, Pan A, Hu FB. Dietary Protein Intake and Risk of Type 2 Diabetes in US Men and Women. Am J Epidemiol. 2016 Apr 15;183(8):715-28. doi: 10.1093/aje/kwv268. Epub 2016 Mar 28. PMID 27022032
- [Background] Song M, Fung TT, Hu FB, Willett WC, Longo VD, Chan AT, Giovannucci EL. Association of Animal and Plant Protein Intake With All-Cause and Cause-Specific Mortality. JAMA Intern Med. 2016 Oct 1;176(10):1453-1463. doi: 10.1001/jamainternmed.2016.4182. PMID 27479196
- [Background] Derbyshire EJ. Flexitarian Diets and Health: A Review of the Evidence-Based Literature. Front Nutr. 2017 Jan 6;3:55. doi: 10.3389/fnut.2016.00055. eCollection 2016. PMID 28111625
- [Background] Edelman M, Colt M. Nutrient Value of Leaf vs. Seed. Front Chem. 2016 Jul 21;4:32. doi: 10.3389/fchem.2016.00032. eCollection 2016. PMID 27493937
- [Background] Rizzo G, Lagana AS, Rapisarda AM, La Ferrera GM, Buscema M, Rossetti P, Nigro A, Muscia V, Valenti G, Sapia F, Sarpietro G, Zigarelli M, Vitale SG. Vitamin B12 among Vegetarians: Status, Assessment and Supplementation. Nutrients. 2016 Nov 29;8(12):767. doi: 10.3390/nu8120767. PMID 27916823